CLINICAL TRIAL: NCT01886547
Title: 2013 Annual National Digital Rectal Exam (DRE) Day: Impact on Prostate Health Awareness and Disease Detection
Brief Title: 2013 Annual National Digital Rectal Exam (DRE) Day Study
Status: Completed | Type: Observational
Sponsor: St. Luke's Medical Center, Philippines (Other)
Collaborators: Philippine Board of Urology (Unknown); Philippine Urology Residents Association (Other)
Responsible Party: Principal Investigator, Michael E. Chua, Head, Continuing Medical Education Committee of Philippine Urological Residents' Association, St. Luke's Medical Center, Philippines
Other Study IDs: PURA-2013
Record Dates: First submitted 2013-06-23; First posted 2013-06-26 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Benign Prostatic Hyperplasia; Prostatitis; Prostate Cancer
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatitis; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- New patient presented with prostate disease: prostate disease identified
  Interventions: Other: Prostate health screening

INTERVENTIONS:
Other: Prostate health screening
  Other Names: Digital rectal examination, International prostate symptoms score quetionnaire

SUMMARY:
We aim to determine the effectiveness of 2013 "Mag paDRE ka" programme in increasing general public awareness on prostate health and promoting prostate health assessment among Filipino males aged 40 or older.

DETAILED DESCRIPTION:
Convenience sampling method will be applied to collect all completed Philippine Urological Association (PUA) survey forms from the 11 Philippine Board of Urology accredited training institutions. A data collection form for the purpose of this study will be used to extract data from the Philippine Urological Association survey forms. The data collection form for this study will extract data, which include basic demographic characteristics of the patients (such as age and educational attainment), family history of prostate cancer, other medical conditions, history of prior prostate screening/ consultation for Lower urinary tract Symptoms or prostate disease. The International Prostate Symptom scores (IPSS) collected will be stratified according to mild (1-7), moderate (8-19) and severe (20-35) and the Filipino version Quality of Life (QoL) ratings will be stratified according to Grade 1, grade 2 and grade 3. DRE findings including the approximation of prostate size and prostate characteristic findings will be clustered to normal in size (20grams or less) versus enlarged (>20grams or 2 fingerbreadths in width), nodular vs non-nodular, doughy or hard, and tender versus non-tender.

Participants will be classified according to the following :

1. Target population for screening or not :

   Target population for screening is defined as Filipino males aged 40 years or older, who also had no previous consultation for Lower urinary tract symptoms (LUTS) or prostate cancer screening in the past 12 months
2. Case Finding for significant LUTS or prostate cancer or not :

Case of LUTS or prostate cancer is defined as Filipino males aged 40 years or older with IPSS > 8, OR, has abnormal Digital rectal exam (DRE) finding, which is defined as nodular OR hard OR tender. However, DRE finding of an enlarged prostate but non-nodular, doughy in character and non-tender will not be considered as a case of LUTS or prostate cancer suspect).

Confidentiality of all data will be assured. The case report forms/ data collection form for this study will not contain any patient identifiers. All patient records will be coded in the electronic database as serial number and PUA-designated Institutional code (i.e. SLMC #0001). Only the investigators of this study and other authorized personnel from PUA will be given access to the study data. The PUA survey forms will be secured, filed and only accessed in PUA secretariat building. The electronic database coded with the data from the data collection from of this study will be set with password, and only the study investigators have access to the password.

ELIGIBILITY:
Inclusion Criteria:

* Filipino male ages 40 or older consulted on "Pa-DRE ka" prostate health screening program 2013
* patients presented to the Philippine Board of Urology accredited 11 training institutions
* Consented for the screening program.
* Completed the questionnaire of International Prostate symptoms score
* Has been examined with digital rectal examination

Exclusion Criteria:

* Patients who have incomplete data and did not consent for the screening program
* Non-Filipino male patients

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Filipino males ages 40 or older
Sampling Method: Non-Probability Sample
Enrollment: 925 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Prostate disease (benign prostatic hyperplasia, prostatitis, Prostate cancer) | 1 year
  number of new diagnosed prostate disease (target population) for Pa-DRE ka day screening program.

SECONDARY OUTCOMES:
Prevalence of Prostate Diseases | 1 year
  total number of patient consulted on Pa-DRE ka day with prostate diseases
International Prostate Symptom Score | 1 year
  Total score of international Prostate Symptoms Score of each patients consulted for Prostate screening program (Pa-DRE ka day)
Prostate gland size estimate | 1 year
  Estimated prostate gland size by digital rectal exam for patients presented to the prostate screening program (Pa-DRE ka day)
Digital rectal examination result | 1 year
  Summary of digital rectal exam findings of patients presented to prostate screening program (Pa-DRE ka day)

CONTACTS AND LOCATIONS:
Locations (1):
- Philippine Urological Association Inc., Quezon City, National Capital Region, Philippines

REFERENCES:
- [Result] Chua ME, Lapitan MC, Morales ML Jr, Roque AB, Domingo JK; Philippine Urological Residents Association (PURA). 2013 Annual National Digital Rectal Exam Day: impact on prostate health awareness and disease detection. Prostate Int. 2014 Mar;2(1):31-6. doi: 10.12954/PI.13039. Epub 2014 Mar 30. PMID 24693532